CLINICAL TRIAL: NCT07107633
Title: A Multicenter, Open-access, Self-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Technetium [99mTc]-H7ND Injection in the Diagnosis of Peritoneal Metastasis of Gastrointestinal Malignancies.
Brief Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of Technetium [99mtc]-H7ND Injection in the Diagnosis of Peritoneal Metastasis of Gastrointestinal Malignant Tumor.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiaxing Pharmadax Genesis Pharmaceutical Technology Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-024R
Record Dates: First submitted 2025-07-10; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor; Peritoneal Metastasis
MeSH Terms: interventions — Technetium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with malignant tumors of the gastrointestinal tract (Experimental)
  Interventions: Drug: Technetium [99mTc]-H7ND injection

INTERVENTIONS:
Drug: Technetium [99mTc]-H7ND injection — Technetium [99mTc]-H7ND injection is a radiolabeled fibroblast activation protein inhibitor

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of technetium [99mTc]-H7ND injection in the diagnosis of peritoneal metastasis of gastrointestinal malignant tumor. Objective: To evaluate the safety of technetium [99mTc]-H7ND injection in the diagnosis of peritoneal metastasis of gastrointestinal malignant tumor. Objective: To explore the diagnostic threshold of technetium [99mTc]-H7ND injection for peritoneal metastasis of gastrointestinal malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

Only those who meet all the following requirements are eligible to join the group:

1. Adults over 18 years of age (based on the time when the informed consent form was signed) can be male or female;
2. Subjects with gastrointestinal malignant tumor confirmed by histology/cytology;
3. Subjects to be surgically removed or explored;
4. The estimated survival time is ≥12 weeks;
5. Subjects of childbearing age agreed to adopt effective contraceptive measures during the study period;
6. Subjects fully understand the purpose, nature, methods and possible adverse reactions of the experiment, voluntarily participate in and sign a written informed consent, and are willing to follow the requirements of the protocol to complete the study.riteria:

Those who meet one of the following items are not allowed to join the group:

1. According to the researcher's judgment, during the screening period, from the imaging examination to the comprehensive real diagnosis information result, the patients were treated with anti-digestive tract tumor;
2. symptomatic brain metastases who need treatment;
3. Have serious cardiovascular and cerebrovascular diseases;
4. There are other contraindications for imaging examination of the research plan, such as claustrophobia;
5. Have a history of other malignant tumors;
6. Pregnant (pregnancy test positive in screening period) or lactating women;
7. Other circumstances that the researcher considers inappropriate to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of technetium [99mTc]-H7ND injection in the diagnosis of peritoneal metastasis of gastrointestinal malignant tumor | 1-7 days from time of injection
  To evaluate whether the sensitivity of 99mTc-H7ND SPECT/CT in the diagnosis of peritoneal metastasis of gastrointestinal malignant tumor is better than that of enhanced CT by SOT.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, China